CLINICAL TRIAL: NCT00622947
Title: The Antidepressant Effect of Right Temporal Kow Frequency rTMS Compared to Sham: A Clinical Controlled, Randomized, Blinded Study
Brief Title: The Antidepressant Effect of Right Temporal Low Frequency rTMS Compared to Sham
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too few patients included
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-20070144
Record Dates: First submitted 2008-01-24; First posted 2008-02-25 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Depressive Disorder
Keywords: Depression; antidepressant effect; rTMS; sham; cognition; saliva cortisol; brain derived neurotropic factor
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- repetitive transcranial magnetic stimulation (Active Comparator): Low frequency ( 1 HZ) rTMS of the right prefrontal cortex. On each of 15 consecutive week days (apart from weekends), the patients received two 60-second1-Hz trains delivered at an intensity of 110% of motor thresholdand with a 180 seconds' intertrain interval.
  Interventions: Procedure: right temporal low frequency (1 hz) rTMS
- Placebo stimulation (Sham Comparator): Sham- rTMS of the right prefrontal cortex. On each of 15 consecutive week days (apart from weekends), the patients received two 60-second1-Hz trains delivered at an intensity of 110% of motor thresholdand with a 180 seconds' intertrain interval.
  Interventions: Procedure: Sham-rTMS

INTERVENTIONS:
Procedure: right temporal low frequency (1 hz) rTMS — Right temporal low frequency (1 hz) rTMS.
  Other Names: A Magstim Rapid stimulator (the Magstim Company Ltd, Whiteland, UK)with a 90 mm circular coil is used.
  Arms: repetitive transcranial magnetic stimulation
Procedure: Sham-rTMS — The coil is angled 90 degrees away from the scalp
  Arms: Placebo stimulation

SUMMARY:
The aim of the present study is to compare the antidepressant effect of low frequency rTMS applied over the right temporal cortex with sham stimulation.

DETAILED DESCRIPTION:
TMS complies focal stimulation of the brain through a time varying magnetic field. Clinical controlled trials indicate that rTMS of the dorsolateral prefrontal cortex may have an antidepressant effect and no serious side effects. Several clinical controlled studies investigating the antidepressant effect of low as well as high frequency rTMS of the right and left prefrontal cortex have been carried out with varying results.Research on the issue suffer from small and selected study populations.There is a need for additional clinical controlled studies on larger samples and methodological investigations to clarify what is the optimal stimulus design for the treatment of depressed patients.

Recent research indicates that Depression is associated with an increased metabolic activity of subcortical areas especially the right hippocampus of the brain.

Remission of depression symptoms is associated with normalisation of the described subcortical hyperactivity.

Low frequency rTMS has shown to be associated with sustained reduction in neuronal activity.

There may be an association between the activity decreasing effect of low frequency rTMS and reduction in psychiatric symptoms.

The investigators want to test the hypothesis that low frequency rTMS of the right temporal subcortical areas (Hippocampus and and the parahippocampal part of CNS) may perform an antidepressant effect by normalizing the described hyperactivity of the subcortical areas in depressed patients.

In addition the investigators want to test whether blood concentration of Brain Derived Neurotropic Factor( BDNF), the BDNF-genotype and saliva cortisol may be of predictive value in depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients admitted to Århus university Hospital , Risskov or outpatients from the psychiatry district centres or practising specialist in the area.
* Moderate - severe depression according to ICD-10/ DSM-IVR
* Age 18-80 years
* Total Hamilton score ( 17-items) of ≥ 18 or subscale score ≥ 9
* Right handed

Exclusion Criteria:

* Organic brain disease
* Epilepsy in growing age
* Metallic objects as the result of a chest or Brain surgery
* Cardiac pacemakers
* Somatic diseases associated with brain dysfunction
* Pregnancy
* Suicide risk of severe degree
* Severe agitation or delirium
* Alcohol and drug dependency
* Ongoing Electroconvulsive treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The total 17-item score on the Hamilton scale for depression | 4 weeks of treatment and 4 weeks of follow-up
  semistructured interview scale.

CONTACTS AND LOCATIONS:
Overall Officials: Poul Erik B Hansen, consultant, Principal Investigator — University Hospital og Aarhus, Denmark
Locations (1):
- University Hospital of Aarhus, Risskov, Aarhus, Risskov, Denmark

REFERENCES:
- [Background] Klein E, Kreinin I, Chistyakov A, Koren D, Mecz L, Marmur S, Ben-Shachar D, Feinsod M. Therapeutic efficacy of right prefrontal slow repetitive transcranial magnetic stimulation in major depression: a double-blind controlled study. Arch Gen Psychiatry. 1999 Apr;56(4):315-20. doi: 10.1001/archpsyc.56.4.315. PMID 10197825